CLINICAL TRIAL: NCT00682149
Title: Effects Polyphenol Containing Antioxidants on Oxidative Stress in Diabetic Patients
Brief Title: Effects of Polyphenol Containing Antioxidants on Oxidative Stress in Diabetic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yeditepe University Hospital (Other)
Responsible Party: Effects of polyphenol containing antioxidants on oxidative stress in type 2 diabetic patients, Yeditepe University Medical Faculty, Family Medicine Department
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DM2-AOC
Record Dates: First submitted 2008-05-20; First posted 2008-05-22 (Estimated); Last update posted 2008-05-22 (Estimated); Status verified 2008-05

CONDITIONS: Type 2 Diabetes
Keywords: Oxidative stress; malondialdehyde; glutathione; diabetes; polyphenol containing antioxidants; diet rich in vegetables; weekly aerobic exercise
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Tea; Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Placebo Comparator): We planned to compare a study group of 60 subjects with a placebo group of 60 subjects
  Interventions: Dietary Supplement: PomGT (500 mg pomegranate extracts, 300 mg green tea and 60mg vitamin C)
- Group 2 (Active Comparator): We planned to compare a study group of 60 subjects with a placebo group of 60 subjects
  Interventions: Dietary Supplement: PomGT (500 mg pomegranate extracts, 300 mg green tea and 60mg vitamin C)

INTERVENTIONS:
Dietary Supplement: PomGT (500 mg pomegranate extracts, 300 mg green tea and 60mg vitamin C) — 1 tablet/day for 3 months
  Other Names: Comilac PomGT tablets

SUMMARY:
There has been an increase in the prevalance of type 2 diabetes in developed countries in recent years. The major contributing factors have been genetic predisposition, environmental factors, and unhealthy eating habits and stress. Adverse effects on cardiovascular and renal systems after prolonged hyperglycemia bring serious burden to patients, to their families and to the society.

Oxidative stress has been defined as the imbalance between the production of reactive oxygen molecules and antioxidant protective molecules. It has been claimed that oxidative stress that the organism is exposed to and disturbance in anti-oxidant mechanisms have been important in the initiation of diabetes and its complications. Malondialdehyde is the final product of lipid peroxidation and it is an aldehyde as well. It has been accepted that malondialdehyde has been a biomarker in measuring oxidative stress.

Type 2 diabetic people who are between 40 -65 years of age will be the subjects of our study. The levels of fasting glucose, HbA1c, LDL, triglyceride, AST and ALT and also malondialdehyte, hydrogen peroxide and oxidative stress will be determined in patients blood after making them consume a 1500 calory standard diet for 2 weeks, The patients will be randomly divided into two grouos at the end of the two weeks. Group 1 will take placebo in addition to the diet, Group 2 will receive polyphenol containing capsules with pomegranate extract (500 mg), green tea extract (300 mg) and a little bit of (60 mg) vitamin C for three months. At the end of three months the measurement of biochemical parameters will be repeated.

Patients with cardiac, renal, liver disease and smokers will be excluded from the study.

Patients in both groups will have a diet rich in vegetables, three servings of fruit, maximum three slices of bread with a total calory of 1500.

In addition to these, both groups will have a weekly aerobic exercise regimen of 150 minutes conducted after breakfast.

The biochemical results of the two groups will be compared at the end of the experiment and they will be statistically evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic patients between 40-65 years of age will be eligible for the study

Exclusion Criteria:

* Patients with cardiac, renal, liver disease and smokers will be excluded from the study.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2008-05; Primary Completion 2008-07 (Estimated); Study Completion 2008-10 (Estimated)

PRIMARY OUTCOMES:
Amelioration of antioxidative capacity in diabetic patients by polyphenol containig antioxidants | 3 months

SECONDARY OUTCOMES:
treatment of type 2 diabetes by polyphenol containing antioxidants | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Aysen Fenercioglu, Assist Prof. Dr., Principal Investigator — Yeditepe University Medical Faculty, Family medicine Department
Locations (1):
- Sisli Etfal Education and Research Hospital, Istanbul, Turkey (Türkiye)